CLINICAL TRIAL: NCT01987492
Title: A Phase II, Randomized, Double-Blind, Placebo Controlled, Multicenter Trial to Assess the Oral Corticosteroid-Sparing Effect of Lebrikizumab in Patients With Severe Corticosteroid Dependent Asthma
Brief Title: A Study of Lebrikizumab (RO5490255) in Participants With Severe Oral Corticosteroids (OCS) Dependent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WB28182; 2012-000190-24 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Lebrikizumab High Dose (Experimental): Participants will receive lebrikizumab at high dose level as subcutaneous (SC) injection every 4 weeks during the 44-week DBPC period, followed by a 32-week ATE period, and during the LTE period.
  Interventions: Drug: Lebrikizumab
- Lebrikizumab Low Dose (Experimental): Participants will receive lebrikizumab at low dose level as SC injection every 4 weeks during the 44-week DBPC period, followed by a 32-week ATE period, and during the LTE period.
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Participants will receive placebo matching to lebrikizumab SC injection every 4 weeks during the 44-week DBPC period. Participants will then be randomized to receive either high- or low-dose lebrikizumab every 4 weeks during the 32-week ATE period and will continue same treatment in the LTE period.
  Interventions: Drug: Lebrikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered as SC injections every 4 weeks at dose and schedule described in arm description.
  Other Names: RO5490255
Drug: Placebo — Placebo matching to lebrikizumab will be administered as SC injections every 4 weeks as per schedule described in arm description.
  Arms: Placebo

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy of lebrikizumab compared with placebo, as measured by the ability of participants to achieve lower daily doses of OCS, among those with severe corticosteroid-dependent asthma. Prednisone/prednisolone will be the OCS therapy prescribed. Participants will be randomized to receive lebrikizumab or matching placebo for 44 weeks in a double-blind, placebo-controlled (DBPC) period. Those who complete the 44-week period may continue into a 32-week active treatment extension (ATE) period, during which all participants will receive lebrikizumab treatment. Following completion of the ATE period, participants who have both tolerated and derived benefit from treatment with lebrikizumab may continue their lebrikizumab treatment into a long-term extension (LTE) period. Participants will transition to 24 weeks of safety follow-up upon discontinuation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma despite intensive follow-up by an asthma specialist for >/=6 months prior to Visit 1
* Baseline forced expiratory volume in 1 second (FEV1) >/=40% of predicted prior to randomization
* Receiving high doses of inhaled glucocorticosteroids at a total daily dose of >/=1500 micrograms (mcg) beclomethasone dipropionate or equivalent and long-acting beta-adrenoceptor agonist (LABA), with or without an additional controller, for at least 3 months prior to Visit 1
* Chronic treatment with maintenance OCS for >/=6 months prior to Visit 1
* Assessment to ensure diagnosis of refractory asthma and OCS dependence on minimal effective or maximum tolerated dose prior to Visit 1 with compliance

Exclusion Criteria:

* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Asthma exacerbation within 28 days prior to Visit 1 or during screening (prior to Visit 3)
* For adults: Active tuberculosis requiring treatment within the 12 months prior to Visit 1
* For adolescents: History of active tuberculosis requiring treatment
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Known current malignancy or current evaluation for a potential malignancy
* History of interstitial lung disease, chronic obstructive pulmonary disease, or other clinically significant lung disease other than asthma
* Infection requiring hospital admission or requiring treatment with intravenous (IV) or intramuscular (IM) antibiotics within 4 weeks prior to Visit 1 or during screening
* Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening
* Active parasitic infection or Listeria monocytogenes infection within 6 months prior to Visit 1 or during screening
* Current smoker or former smoker with a smoking history of more than 15 pack-years
* Current use of an immunomodulatory/ immunosuppressive therapy or past use within 3 months or 5 drug half-lives (whichever is longer) prior to Visit 1
* Use of a licensed or investigational monoclonal antibody other than anti-interleukin (IL)-13 or anti-IL-4/IL-13, including but not limited to, omalizumab, anti-IL-5, or anti-IL-17, within 6 months or 5 drug half-lives (whichever is longer) prior to Visit 1
* Receipt of a live attenuated vaccine within the 4 weeks prior to Visit 1 during screening or anticipation of receipt of a live attenuated vaccine throughout the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Relative Change From Baseline in Daily OCS Dose at Week 44 | Baseline, Week 44

SECONDARY OUTCOMES:
Absolute Change From Baseline in Daily OCS Dose at Week 44 | Baseline, Week 44
Relative Change From Week 12 in Average OCS Dose at Week 44 | Week 12, Week 44
Percentage of Participants Achieving at Least a 50 percent (%) Reduction in Their Daily OCS Dose at Week 44 Relative to Baseline | Baseline, Week 44
Percentage of Participants Discontinuing OCS Therapy or Having Achieved an Adrenal Maintenance Dose at Week 44 | Week 44
  Percentage of participants discontinuing OCS therapy or having achieved adrenal maintenance dose (cortisol level less than or equal to 100 nanomoles per liter) will be reported.
Percentage of Participants With Asthma Exacerbations | Baseline up to Week 44
  An asthma exacerbation is defined as new or increased asthma symptoms (including wheeze, cough, dyspnea, chest tightness, or nocturnal awakenings due to these symptoms) that lead to treatment with systemic corticosteroids greater than or equal to (>/=) 30 milligrams (mg) or 0.5 mg per kilogram (kg) for >/=3 consecutive days or to hospitalization.
Percentage of Participants With Adverse Events | Baseline up to 24 weeks after last dose administration (up to a minimum of approximately 2 years)
Percentage of Participants With Anti-therapeutic Antibodies (ATAs) Against Lebrikizumab | Predose (0 hours) at Weeks 0, 4, 12, 24, 36, 44, 52, 64, and 76, at early discontinuation (up to a minimum of approximately 2 years), and at 24 weeks after last dose administration (up to a minimum of approximately 2 years)
Minimum Observed Serum Lebrikizumab Concentration (Cmin) | Predose (0 hours) at Weeks 4, 12, 24, 36, and 44

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (71):
- United States (9):
  - Kern Allergy Med Clinic, Inc., Bakersfield, California
  - Allergy & Asthma Care Center of Southern California, Long Beach, California
  - South Florida Research Center, Inc., Miami, Florida
  - Georgia Pollens, Albany, Georgia
  - Mount Sinai Medical Center, New York, New York
  - Allergy & Immunology, Tulsa, Oklahoma
  - Pioneer Research Solutions, Houston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Pulmonary Consultants PLLC, Tacoma, Washington
- Australia (3):
  - Princess Alexandra Hospital, Department of Respiratory and Sleep Medicine, Brisbane, Queensland
  - Monash Medical Centre; Respiratory and Sleep Medicine, Clayton, Victoria
  - Institute for Respiratory Health Inc, Nedlands, Western Australia
- Belgium (3):
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - Longartsenpraktijk, Genk
  - UZ Gent, Ghent
- Inspiration Research Limited, Toronto, Ontario, Canada
- Czechia (4):
  - Hornmed, Brno
  - Nemocnice Liberec; KNL a.s. - TRN, Liberec
  - Nemocnice Nový Jičín, Nový Jičín
  - Rokycanska nemocnice, Rokycany
- Gentofte Hospital, Klinik for Allergi, Hellerup, Denmark
- France (9):
  - CHU de Grenoble - Hôpital André Michallon, Grenoble
  - CH de Bicetre; Pneumologie, Le Kremlin-Bicêtre
  - Hôpital de La Croix Rousse, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes - Hôpital Laennec; Service de Pneumologie, Nantes
  - CHU de Nice, Nice
  - Hopital Bichat Claude Bernard ; Service de Pneumologie, Paris
  - CHU de Haut Leveque, Pessac
  - Nouvel Hôpital Civil; Pôle de Pathologie Thoracique, Strabourg
- Mexico (3):
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Centro Investigacion Medico Biologica y Terapia Avanzada, Guadalajara
  - Centro Integral Médico SJR SC, Querétaro
- Netherlands (3):
  - Academisch Medisch Centrum; Afdeling Longziekten, F5-258, Amsterdam
  - Spaarne Ziekenhuis Hoofddorp; Long Geneeskunde, Hoofddorp
  - Antonius Ziekenhuis; Dept of Lung Diseases, Nieuwegein
- New Zealand (4):
  - NZ Respiratory & Sleep Institute, Auckland
  - Dunedin Hospital, Dunedin
  - Clinical Trials Unit, Bay of Plenty District Health Board, Tauranga
  - Medical Research Inst. of New Zealand; Respiratory, Wellington
- Poland (7):
  - Specjalistyczny Osrodek Alergologiczno-Internistyczny ALL-MED, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Specjalistyczna Poradnia Pulmonologiczna, Ostrów Wielkopolski
  - Niepubliczny Zaklad Opieki Zdrowotnej PROFILAKTYKA Wladyslaw Pierzchala, Ruda Śląska
  - Klinika Chorób Wewnetrznych i Alergologii MSW, Warsaw
  - EMC Instytut Medyczny SA; Przychodnia przy ulicy Łowieckiej, Wroclaw
- Puerto Rico (2):
  - San Juan Bautista School of Medicine-Clinical Research Unit, Caguas
  - Advanced Medical Concepts, PSC, Cidra
- Slovakia (2):
  - ZAPA JJ Sro, Levice
  - Plucna ambulancia, Spišská Nová Ves
- University Clinic of Pulmonary and Allergic Diseases Golnik, Golnik, Slovenia
- Spain (5):
  - Complejo Hospitalario Universitario de Santiago; Servicio de Neumología, Santiago de Compostela, La Coruña
  - Hospital de la Santa Creu; i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario de Salamanca; Servicio de Neumologia, Salamanca
  - Hospital Universitario Doctor Peset, Valencia
- United Kingdom (14):
  - Belfast City Hospital; Respiratory Department, Belfast
  - Heartlands Hospital; Respiratory Department, Birmingham
  - Gartnavel General Hospital; Respiratory Department, Glasgow
  - New Lister Buliding, Level 1; Clinical Research Facility, Glasgow
  - Royal Hospital For Children, Glasgow
  - Southampton General Hospital; Respiratory Department, Hampshire
  - Leicester Royal Infirmary NHS Trust, Leicester
  - Glenfield Hospital; Respiratory -Allergy Unit, Leicester
  - St Bartholomew's Hospital (Barts); Respiratory Department, London
  - Royal Brompton Hospital; Respiratory Department, London
  - Wythenshawe Hospital; North West Lung Research Centre, Manchester
  - Freeman Hospital; Respiratory Department, Newcastle upon Tyne
  - Derriford Hospital; The Lind Research Department, Plymouth
  - Sheffield Clinical Research Facility; National Institute for Health Research, Sheffield